CLINICAL TRIAL: NCT00788216
Title: Development and Validation of A Comprehensive Instrument to Determine Utilities for Health States Relevant to Cervical Gynecologic Cancer Patients
Brief Title: Development & Validation of Utilities for Health States Relevant to Cervical Cancer Patients
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00008129
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Cancer
Keywords: Radical hysterectomy; Whole pelvic radiation; Brachytherapy; Chemoradiation; Complications; Quality of Life
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Women over the age of 18 without the diagnosis of cervical cancer.
  Interventions: Other: Discussion & scoring of health states related to the treatment of cervical cancer
- Cervical Cancer Patients: Women over the age of 18 with a history of cervical cancer treated with surgery or chemoradiation.
  Interventions: Other: Discussion & scoring of health states related to the treatment of cervical cancer

INTERVENTIONS:
Other: Discussion & scoring of health states related to the treatment of cervical cancer — Subjects will be interviewed using the visual analog score and time trade off methods.
  Other Names: Ultities Scores

SUMMARY:
Purposes of this study: 1) To define comprehensive set of descriptive health states related to treatment of cervical cancer (e.g. radical hysterectomy, whole pelvic radiation, brachytherapy, chemoradiation) 2) To define set of descriptive health states related to adverse events associated w treatment of cervical cancer (i.e. bladder dysfunction, pain, enteritis, fistula formation) & 3) To derive, using a validated method, a set of QoL related utility scores corresponding to these health states.

DETAILED DESCRIPTION:
Subjects will valuate cervical cancer-related health states using the visual analog score (VAS) and TTO (TTO) methods. The subject will be asked to read a pertinent health state description and listen while it is read aloud. She will first be asked to place the state on a continuum (VAS) from zero to 100, with 100 presenting perfect health and zero presenting death. The TTO interview will then be administered. The subject will be asked to assume a remaining life expectancy of 30 years, and to choose between 30 years in the health state described or 29 years in a state of perfect health. The utility of the health state, a number between zero and one, is calculated as the minimum number of years the patient would accept divided by 30. Each subject will be asked to review and valuate 20 health states over the course of 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Any member of public over age of 18 and without the diagnosis of cervical cancer can participate in this study.
* Patients over the age of 18 with the diagnosis of cervical cancer are eligible to participate in this study.

Exclusion Criteria:

* Any member of public under the age of 18 or with a prior diagnosis of cervical cancer is excluded from this study.
* Any cervical cancer patient younger than 18 is excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the Public- Members of the public are considered the standard group to assign utilities for health-economic purposes. Forty-five members of the public, without a diagnosis of cervical cancer, will be recruited.
  Cervical Cancer Patients- Fifteen patients, with a diagnosis of cervical cancer (either currently being treated or previously treated).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The development and validation of a comprehensive set of quality of life related utility scores for the treatment of cervical cancer. | lifetime

SECONDARY OUTCOMES:
To incorporate these utility scores into a previous decision model which will allow for outcomes, costs, and quality of life to be analyzed in the treatment of cervical cancer patients. | lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Havrilesky, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States